CLINICAL TRIAL: NCT00336908
Title: Inflammatory Responses of Intravenous Fish Oil, Soybean Oil and Medium Chain Triglyceride Fat Emulsions in Young Children Before and After Open Heart Surgery
Brief Title: Inflammatory Responses to Lipid Emulsions in Children Before and After Open Heart Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Stollery Children's Hospital Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2030001 71860000074; UofA-JVA-2005-1
Record Dates: First submitted 2006-06-13; First posted 2006-06-14 (Estimated); Last update posted 2007-11-27 (Estimated); Status verified 2007-11

CONDITIONS: Inflammation; Cardiac Surgical Procedures
Keywords: Intensive Care,Neonatal; Parenteral nutrition; Fat emulsions,Intravenous
MeSH Terms: conditions — Inflammation; Hyperphagia | interventions — Fish Oils

INTERVENTIONS:
Drug: a combination of MCT, LCT , and Fish Oil

SUMMARY:
This study is a blinded, randomized, controlled prospective trial comparing immune response (sepsis, inflammatory response, pulmonary vasoconstriction) in 2 groups of infants less than 3-month old receiving pre and post cardiopulmonary bypass surgery. The infants will receive 1 out of the 2 following intravenous lipid preparations: Soybean Oil (n-6), or a combination of Medium Chain Triglyceride i.e. coconut oil, Long Chain Triglyceride i.e. Soybean Oil, and Fish Oil (MCT:LCT:FO). There will be 16 subjects in each group.

ELIGIBILITY:
Inclusion Criteria:

* 36 weeks gestation
* 3 months corrected age
* appropriate for gestational age (AGA)
* admitted for surgical correction of congenital heart defects (single ventricle, tetralogy of Fallot, truncus and complex biventricular repairs)
* enteral nutrition at 30 kcal/kilogram/day

Exclusion Criteria:

* 5 minute Apgar score of 4
* major congenital defect other than heart defect
* presence of significant neonatal morbidity (intraventricular hemorrhage (IVH) grade 3 or greater, necrotizing enterocolitis (NEC) and surgical abdomen)
* any metabolic disorder
* any endocrine disorder
* medications which alter eicosanoid metabolism including indomethacin, acetylsalicylate (with exception of steroids which will be analyzed independently)

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Estimated)
Dates: Start 2005-11; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
To determine whether incidence of sepsis and degree of inflammatory response is altered

SECONDARY OUTCOMES:
To characterize serum arachidonic acid and eicosapentaenoic acid levels, leukotriene B 4/leukotriene B 5 levels and incidence of nosocomial infection
To characterize incidental findings as a result of attaining complete fatty acid and cytokine profiles

CONTACTS AND LOCATIONS:
Overall Officials: John E Van Aerde, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] Larsen BM, Goonewardene LA, Joffe AR, Van Aerde JE, Field CJ, Olstad DL, Clandinin MT. Pre-treatment with an intravenous lipid emulsion containing fish oil (eicosapentaenoic and docosahexaenoic acid) decreases inflammatory markers after open-heart surgery in infants: a randomized, controlled trial. Clin Nutr. 2012 Jun;31(3):322-9. doi: 10.1016/j.clnu.2011.11.006. Epub 2011 Dec 3. PMID 22136963